CLINICAL TRIAL: NCT07265674
Title: A Phase 3, Multicenter, Randomized, Open-label, Study Evaluating the Efficacy and Safety of Nanvuranlat in Patients With Previously Treated Advanced Biliary Tract Cancer
Brief Title: A Study to Select a Dose Regimen (Part A) and to Investigate Overall Survival (Part B) With Nanvuranlat Compared With Physician's Best Choice in Participants Aged 18 Years or Older With Biliary Tract Cancer
Acronym: Beacon-BTC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: J-Pharma Co., Ltd. (Industry)
Collaborators: Uniphar Development, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JPH203-P3-BTC
Record Dates: First submitted 2025-11-11; First posted 2025-12-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Advanced Biliary Tract Cancer; Biliary Tract Cancer (BTC)
Keywords: Intrahepatic cholangiocarcinoma (IHC); Extrahepatic cholangiocarcinoma (EHC); Gallbladder carcinoma (GBC)
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms | interventions — Folfox protocol; Leucovorin; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Nanvuranlat 50mg (Experimental): Nanvuranlat 50mg administered via a 90-minute intravenous infusion once daily for 5 consecutive days, followed by 9 days off treatment
  Interventions: Drug: Nanvuranlat
- Navuranlat 75mg (Experimental): Nanvuranlat 75mg administered via a 90-minute intravenous infusion once daily for 5 consecutive days, followed by 9 days off treatment
  Interventions: Drug: Nanvuranlat
- Navuranlat 375mg (Experimental): Nanvuranlat 375mg administered via a 46-hour continuous intravenous infusion once every 14 days
  Interventions: Drug: Nanvuranlat
- Physicians Best Choice (PBC) (Other): 1. FOLFOX regimen (Leucovorin, 5-Flurouracil and Oxaliplatin) administered on Day 1 of each 14 day cycle, or
  2. FOLFIRI regimen (Leucovorin, 5-Flurouracil and Irinotecan) administered once during 14 day cycle, or
  3. Best Supportive Care (BSC) including symptomatic therapeutics, palliative radiation for pre-existing metastases and transfusion of blood products administered at discretion of Investigator.
  Interventions: Other: Physician's Best Choice

INTERVENTIONS:
Drug: Nanvuranlat — Nanvuranlat, IV administration
  Arms: Nanvuranlat 50mg; Navuranlat 375mg; Navuranlat 75mg
Other: Physician's Best Choice — 1. FOLFOX regimen (Leucovorin, 5-Flurouracil and Oxaliplatin) administered on Day 1 of each 14 day cycle, or
  2. FOLFIRI regimen (Leucovorin, 5-Flurouracil and Irinotecan) administered once during 14 day cycle, or
  3. Best Supportive Care (BSC) including symptomatic therapeutics, palliative radiation for pre-existing metastases and transfusion of blood products administered at discretion of Investigator.
  Other Names: FOLFOX Regimen (Leucovorin, 5-Flurouracil and Oxaliplatin; FOLFIRI Regimen (Leucovorin, 5-Flurouracil and Irinotecan); Best Supportive Care (BSC)
  Arms: Physicians Best Choice (PBC)

SUMMARY:
This study is designed to 1) select a dose regimen for continued development and 2) evaluate nanvuranlat versus Physicians Best Choice (PBC) (FOLFOX, FOLFIRI, or Best Supportive Care (BSC)) in participants aged 18 years and over with BTC. Participants enrolling in Part A the trial will be randomly assigned to receive 1 of 3 nanvuranlat dose regimens or PBC. In Part B, participants will be randomly assigned to receive nanvuranlat or PBC. Participants will receive treatment every 2 weeks for as long as they do not experience safety issues, or their cancer gets worse, and the study doctor feels they should stop treatment. Health measurements including physical examinations, vital signs, ECGs, and safety laboratory tests will be performed to monitor safety, and tumor imaging will be performed to monitor cancer response to treatment. Other exploratory makers will be measured to better understand how nanvuranlat works.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, open-label, 2-part study designed to select a dose regimen for continued development (Part A) and evaluate the efficacy and safety of nanvuranlat versus PBC (Part B) for the treatment of patients with advanced (locally advanced or metastatic) BTC who have previously received 1 prior standard therapy for advanced BTC plus appropriate therapies targeting druggable molecular mutations/aberrations. Randomization will be stratified by disease subtypes: IHC, EHC, and GBC.

Part A (Dose Regimen Selection) - Three nanvuranlat dose regimens will be evaluated in Part A. Cohorts 1 and 2 will receive 50 or 75 mg of nanvuranlat via a 90-minute infusion, once daily for 5 days, followed by 9 days treatment free (Nanvuranlat-5/9). Cohort 3 will receive 375 mg of nanvuranlat via a 46-hour infusion once every 14 days (Nanvuranlat-46). Participants will be randomized 1:1:1:1 to 4 cohorts. Each treatment cycle will be 14 days and study intervention will be administered beginning on Day 1 during each treatment cycle, except for those participants receiving BSC who will receive care at the discretion of the Investigator.

Part B (Efficacy Evaluation) - Participants will be randomized 1:1 to either nanvuranlat (dose regimen selected in Part A) or PBC (FOLFOX, FOLFIRI, or BSC). Each treatment cycle will be 14 days and study intervention will be administered beginning on Day 1 during each treatment cycle, except for those participants receiving BSC who will receive care at the discretion of the Investigator.

ELIGIBILITY:
Inclusion Criteria:

- Individuals are eligible to be included in the study only if all of the following criteria apply:

1. At least 18 years of age inclusive at the time of signing the informed consent.
2. Provides informed written consent according to local laws or regulations.
3. Able and willing to comply with scheduled visits, treatment plans, procedures, and laboratory tests, including peripheral blood and urine sampling during the study.
4. Willing to participate in LAT1 testing and NAT2 and transporter genotyping. Note: For LAT1 testing, if the participant does not have archival tissue and a fresh biopsy is not in the best interest of the participant, they will still be eligible for the trial.
5. Cancer must be metastatic, locally advanced and unresectable, or not amenable to treatment with local therapies that could offer a reasonable likelihood of clinical benefit.
6. Histologic or cytologic diagnosis of BTC.
7. Has BTC that is classified as either an IHC, EHC, or GBC based on surgical, clinical, or laparoscopic findings and/or radiological imaging (eg, CT, MRI).
8. Has received 1 prior appropriate platinum (cisplatin, carboplatin, or oxaliplatin)-based therapy for advanced disease (locally advanced or metastatic) with or without a mAb targeting PD-1 or PD-L1.

   1. Disease progression during or within 6 months of neoadjuvant or adjuvant treatment with a platinum-containing regimen will count as having received 1 prior regimen.
   2. If a patient has a mutation/fusion of IDH1, FGFR2 or NTRK, or an amplified, mutated, or overexpressed form of HER2, or a recognized aberration in a validated "driver" of BTC, and was treated with an appropriate targeted agent, or the patient's tumor was determined to be MSI-H and an appropriate PD-1/PD-L1 mAb was administered, the targeted therapy or immunotherapy will NOT count as a separate line of treatment.
9. ECOG PS of 0 or 1.
10. Expected life expectancy of at least 90 days after the first day of treatment as per the site Investigator.
11. At least 1 measurable lesion by RECIST v1.1 based on imaging (eg, CT, MRI) performed within 28 days prior to initiation of study intervention. Those who have received prior local therapy, including but not limited to embolization, chemoembolization, radiation therapy, and/or other appropriate ablative procedures to a measurable lesion that is within the treatment and shown ≥ 20% growth in size since posttreatment assessment.
12. Resolution to ≤ Grade 1 by the NCI CTCAE v 5.0 (or higher) of all clinically significant toxic effects of prior chemotherapy or other treatments, except for alopecia and peripheral neuropathy (these must have resolved to ≤ Grade 2). If medical therapy is required for the treatment of a laboratory abnormality, the dose and laboratory value(s) should be stable.
13. Adequate hematologic function:

    1. ANC ≥ 1.5 × 109/L. Myeloid growth factors must not have been administered within 7 days before the participant's first dose of study intervention.
    2. Hemoglobin ≥ 8.5 g/dL and no RBC transfusions during the 14 days before the participant's first dose of study intervention.
    3. Platelet count ≥ 100 × 109/L and no platelet transfusions during the 14 days before the participant's first dose of study intervention.
14. Adequate baseline organ function, as demonstrated by the following:

    1. eGFR ≥ 50 mL/min as estimated by CKD-EPI 2021.
    2. Bilirubin ≤ 2 × ULN (local institution).
    3. AST and ALT ≤ 5 × ULN (local institution).
15. Adequate coagulation function as defined by INR ≤ 1.5 OR a PT ≤ 1.5 × ULN AND an aPTT ≤ 1.5 × ULN if not receiving anticoagulation therapy. Note: Participants may receive subtherapeutic doses of warfarin while on study to maintain patency of venous devices but not with therapeutic doses of warfarin. Participants may be treated with low-molecular weight heparin.
16. Women of childbearing potential must be willing to use a highly effective method of contraception throughout the study and study follow up or for at least 9 months after the last dose of study intervention. Note: A woman is of nonchildbearing potential if she meets 1 of the following criteria: a) postmenopausal with at least 12 months of spontaneous amenorrhea; b) has had a bilateral oophorectomy; or c) has had a hysterectomy. Highly effective methods of contraception include:

    * Abstinence from sexual activity.
    * Hormonal contraception (eg, injection, implant, pill, patch, or vaginal ring as available in each country) associated with inhibition of ovulation (both estrogen and progestogen and progestogen only) in use for at least 30 days before administration of study intervention.
    * Intrauterine device in use for at least 30 days before administration of study intervention.
    * Intrauterine hormone-releasing system in use for at least 30 days before administration of study intervention.
    * Bilateral tubal occlusion/ligation at least 6 months before administration of study intervention.
    * Partner who has been vasectomized at least 6 months before administration of study intervention.
17. Males and their female partners must use a highly effective method of birth control if female partner(s) is of childbearing potential, and males must not donate sperm during the study and for 9 months after the last dose of study intervention.

Exclusion Criteria:

* Individuals will be excluded from study participation if they meet any of the following criteria:

  1. Received systemic therapy or an investigational agent before washing out, as follows:

     1. < 2 weeks prior to Cycle 1 Day 1 for systemic non-immune-based therapy
     2. < 3 weeks prior to Cycle 1 Day 1 for immune-based therapy
     3. ≤ 5 half-lives or 3 weeks (whichever is longer) prior to Cycle 1 Day 1 for an investigational agent
  2. Received radiotherapy to metastatic sites within 2 weeks of Cycle 1 Day 1. Patients must have recovered from all radiation-related toxicities and not require corticosteroids. A 1 week washout is permitted for palliative radiation with a limited port ≤ 2 weeks of radiotherapy to non-CNS disease.
  3. Underwent hepatic radiation, chemoembolization, or radiofrequency ablation < 4 weeks prior to Cycle 1 Day 1.
  4. Underwent major surgery < 3 weeks before Screening and has not recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention.
  5. Known active CNS metastases and/or carcinomatous meningitis. Those with previously treated brain metastases may participate provided they are radiologically stable (ie, without evidence of PD for at least 4 weeks by repeat imaging), clinically stable, and without requirement of corticosteroid treatment for at least 14 days prior to first dose of study intervention. For those with a history of CNS involvement, repeat imaging should be performed during study screening. However, CNS imaging is not required prior to study entry unless there is clinical suspicion of CNS involvement.
  6. Clinically significant cardiovascular disease (eg, uncontrolled or any New York Heart Association Class 3 or 4 heart failure, uncontrolled angina, history of myocardial infarction, unstable angina, or stroke within 6 months prior to study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication).
  7. Resting QTcF > 470 msec at screening.
  8. An additional active malignancy that is progressing or has required active treatment within the past 3 years. Cases involving a past cancer history with substantial potential for recurrence must be discussed with the Medical Monitor before study entry. Patients with the following concomitant neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ (including transitional cell carcinoma, cervical intraepithelial neoplasia, breast cancer, and melanoma in situ), organ-confined prostate cancer with no evidence of PD.
  9. Require strong inhibitors of P-gp, BCRP, OATP1B1, OATP1B3, OATP1A2, and OAT3 transporters unless they can be transferred to other medications within ≥ 5 half-lives of treatment.
  10. Require sensitive substrates of OATP1B1 and OATP1B3 unless they can be transferred to other medications within ≥ 5 half-lives of treatment.
  11. Known positive status for HIV, has not been treated with established appropriate antiretroviral therapy for at least 4 weeks, and has a hydrophobic interaction chromatography viral load < 400 copies/mL and a CD4+ T-cell (CD4+) counts ≥ 350 cells/µL prior to enrollment. No HIV testing is required unless mandated by local health authority.
  12. Active or chronic HBV and active (not cured) HCV. Participants who are HBV carriers without active disease (HBV DNA titer < 1000 copies/mL or 200 IU/mL) or cured HCV (negative HCV RNA test) with confirmed viral clearance that are not receiving ongoing treatment and without residual chronic liver disease may be enrolled.
  13. An uncontrolled intercurrent illness including, but not limited to medical illness; uncontrolled infection requiring therapy; psychiatric illness; alcohol or drug dependence; social situations or a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating Investigator or Medical Monitor.
  14. Requires therapeutic doses of warfarin (ie, requires monitoring). A washout period of 7 days before administration of a participant's first dose of study intervention is required for those in whom therapeutic doses of warfarin are discontinued. Note: Warfarin at a low daily dose to maintain patency for indwelling venous catheters is allowed. Low-molecular weight heparin and direct-acting oral anticoagulants, according to the inclusion requirements pertaining to coagulation test results, are allowed.
  15. Clinically significant edema or intracavitary fluid collections (eg, ascites, pleural effusion, pericardial effusions) resulting in moderate symptoms and/or requiring frequent drainage.
  16. Previously developed shock, anaphylaxis, or renal disorder due to SBECD.
  17. WOCBP who is pregnant, lactating, or discontinued lactation < 12 weeks prior to Screening, or who plans to become pregnant or initiate lactation during the study.
  18. Known reaction or contraindication to any component of study intervention (ie, oxaliplatin, leucovorin [including levoleucovorin], and 5-FU [FOLFOX] and irinotecan, leucovorin, and 5-FU [FOLFIRI]).
  19. Known DPD deficiency. Screening for DPD deficiency is not mandated but should be considered in subjects who have had severe toxicity due to fluoropyrimidine-based therapy in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Part A: Preliminary Overall Survival (OS) | From date of first dose of study intervention until death [Approx. 24 months].
  OS is defined as the time from the date of Cycle 1 Day 1 to the date of death from any cause.
Part B: Overall Survival | From date of first dose of study intervention until death [Approx. 36 months]
  OS is defined as the time from the date of Cycle 1 Day 1 to the date of death from any cause.

SECONDARY OUTCOMES:
Part B: Progression Free Survival | From first dose of study intervention until disease progression or death (which ever occurs first) [Approx. 36 months].
  PFS is defined as the time from the date of Cycle 1 Day 1 to the date of objectively determined progression of disease per the Investigators using RECIST version 1.1 or death from any cause, whichever occurs first.
Part B: Objective Response Rate | From first dose of study intervention until disease progression or death (which ever occurs first) [Approx. 36 months].
  ORR, defined as the proportion of patients achieving a best response of CR or PR per the Investigators using RECIST version 1.1.
Part B: Incidence of treatment-emergent adverse events (TEAEs) | From first dose of study intervention and up to 30 days after last dose of study intervention [Approx. 36 months].
  Incidence of TEAEs, including serious adverse events (SAEs)
Part B: Relative Dose Intensity | From first dose of study intervention and up to first 8 weeks of treatment [Approx. 36 months].
  Relative dose intensity is defined as the ratio of completed infusions to the total planned infusions of the study drug during the first 8 weeks of treatment.
Part B: Dose Reductions, Interruptions and Discontinuations | From first dose of study intervention through last dose of study drug intervention [Approx. 36 months].
  Incidence of dose reductions, Interruptions and Discontinuations
Part B: Electrocardiograms | From first dose of study intervention through last dose of study drug intervention [Approx. 36 months].
  Proportion of patients with treatment-emergent clinically significant ECG abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Eric K Rowinsky, MD, Study Director — Uniphar Development, LLC; Ghassan Abou-Alfa, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (18):
- United States (18):
  - Banner MD Anderson Cancer Center (Site 106), Gilbert, Arizona
  - City of Hope (Site 107), Duarte, California
  - University of California at Irvine (Site 101), Orange, California
  - UCLA Medical Center (Site 117), Santa Monica, California
  - Norton Cancer Institute (Site 115), Louisville, Kentucky
  - Ochsner Medical Center (Site 120), New Orleans, Louisiana
  - Henry Ford Cancer Center (Site 113), Detroit, Michigan
  - Karmanos Cancer Center (Site 109), Detroit, Michigan
  - Masonic Cancer Center, University of Minnesota (Site 116), Minneapolis, Minnesota
  - Rutgers Cancer Institute of New Jersey (Site 103), New Brunswick, New Jersey
  - Rosewell Park Comprehensive Cancer Center (Site 114), Buffalo, New York
  - Memorial Sloan Kettering Cancer Center (Site 108), New York, New York
  - University Hospitals Cleveland Medical Center Seidman Cancer Center (Site 111), Cleveland, Ohio
  - James Cancer Hospital and Solove Research Institute (Site 119), Columbus, Ohio
  - Mercy Clinic (Site 110), Oklahoma City, Oklahoma
  - Allegheny Health Network (Site 121), Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center (Site 104), Dallas, Texas
  - University of Texas MD Anderson Cancer Center (Site 102), Hosuton, Texas

IPD SHARING:
Plan to Share IPD: Undecided
A decision on the sharing of IPD will be made upon completion of Part A (Dose Selection) of the study.

REFERENCES:
- [Background] Furuse J, Ikeda M, Ueno M, Furukawa M, Morizane C, Takehara T, Nishina T, Todaka A, Okano N, Hara K, Nakai Y, Ohkawa K, Sasaki T, Sugimori K, Yokoyama N, Yamamoto K. A Phase II Placebo-Controlled Study of the Effect and Safety of Nanvuranlat in Patients with Advanced Biliary Tract Cancers Previously Treated by Systemic Chemotherapy. Clin Cancer Res. 2024 Sep 13;30(18):3990-3995. doi: 10.1158/1078-0432.CCR-24-0461. PMID 39058429
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39058429/